CLINICAL TRIAL: NCT00922727
Title: Phase I Safety and Tolerance of Lactobacillus Reuteri in Adults
Brief Title: Safety of Lactobacillus Reuteri (L. Reuteri) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, J. Marc Rhoads, Director of Pediatric Gastroenterology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-MSC-08-0266; R21AT003519-01A2 (NIH); U01AT003519 (NIH)
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Colic; Gastrointestinal Tract Infections
Keywords: L. reuteri; Cytokines; Toll like receptors; Healthy Adults; Probiotics
MeSH Terms: conditions — Colic | interventions — Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L. reuteri (Active Comparator): Lactobacillus reuteri oil drops are a natural product containing Lactobacillus reuteri (LR), which has traditionally been used for the establishment and maintenance of a well-functioning gastro-intestinal (GI) tract microflora and prevention and treatment of mild diarrhea associated with GI-tract infections, travel or antibiotic treatment. The oil drops contain a dietary supplement of Lactobacillus reuteri DSM 17938.
  Interventions: Biological: L. reuteri
- Sunflower Oil (Placebo Comparator): Placebo will be the equivalent number of drops of suspended sunflower oil (without LR), provided by Biogaia.
  Interventions: Biological: Sunflower Oil

INTERVENTIONS:
Biological: L. reuteri — The oil drops contains 10^8 CFU (colony forming units). As suggested by the manufacturer in the Certificate of Analysis the daily dose given to each patient will be 5 x 10^8 CFU/ 5 drops. The dose given is within the release limit which is greater than 2 x 10^8 CFU/ 5 drops and less than 8 x 10^8 CFU/ 5 drops.
  Other Names: BioGaia Drops
  Arms: L. reuteri
Biological: Sunflower Oil — As suggested by the manufacturer in the Certificate of Analysis the daily dose given to each patient will be 5 x 10^8 CFU/ 5 drops.
  Other Names: Placebo
  Arms: Sunflower Oil

SUMMARY:
This study will evaluate the safety and tolerability of the probiotic Lactobacillus reuteri (LR) in healthy adult patients. Patients will be randomized to receive either LR or placebo orally each day for a total of 60 doses. The effects on fecal bacteria, circulating white blood cell receptors and inflammatory cytokine profiles will be measured.

DETAILED DESCRIPTION:
Lactobacillus reuteri oil drops are a natural product containing Lactobacillus reuteri (LR), which has traditionally been used for the establishment and maintenance of a well-functioning gastro-intestinal (GI) tract micro flora and prevention and treatment of mild diarrhea associated with GI-tract infections. The oil drops contain a dietary supplement of Lactobacillus reuteri DSM 17938. The patients will receive 5 drops (10^8 live organisms) by mouth daily for 60 days. Daily administration will include 5 drops (5x10^8) of L. reuteri or placebo daily for two months. During this time,circulating peripheral blood mononuclear cell (PBMC) toll-like receptor-2 and -4 levels will be measured, along with PBMC cytokine production levels in vitro. Fecal DGGE analysis(with sequencing of bacterial rDNA) will be completed identifying changes in fecal microbiota. Inflammation in the gut will also be assessed by fecal calprotectin assay (ELISA). The time on study treatment is 2 months, with 4 months observation, for a total of 6 months. There will be 7 required visits, during which, we will assess safety and immune system effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults (18 - 60 years old)
* No other recognized illness

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patient taking immunosuppressive medications, including oral corticosteroids
* Positive result of HIV, Hepatitis B, and/or Hepatitis C test
* Abnormal lab test results
* Gastrointestinal related diseases and surgeries
* Patients with an allergy to antibiotics
* Presence of fever or a pre-existing adverse event monitored in the study
* No more than two study participants in one household
* Use of probiotics in the last 90 days
* Diarrheal illness within the past 30 days
* Recent or current use of oral antibiotics /anti-fungals(in the past 2 weeks)
* Current use of oral laxatives
* Chronic alcohol use or more than 1 drink per day
* Subjects with implanted prosthetic devices including prosthetic heart valves
* Known sensitivity to sunflower oil or products containing linolenic/oleic acids
* Will require that subject not take any other probiotic-containing products, including yogurt supplemented with probiotics during the 6-month period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Treatment of adults with probiotic (health-promoting bacteria) LR, will be safe and well-tolerated. | 8/1/2009 - 7/1/2009

SECONDARY OUTCOMES:
Determine if LR treatment affects circulating levels of pro-inflammatory and anti-inflammatory cytokines, along with expression levels of toll like receptors (TLRs)-2 and -4 in circulating peripheral blood mononuclear cells. | 4/1/2009-7/1/2009

CONTACTS AND LOCATIONS:
Overall Officials: J. Marc Rhoads, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Mangalat N, Liu Y, Fatheree NY, Ferris MJ, Van Arsdall MR, Chen Z, Rahbar MH, Gleason WA, Norori J, Tran DQ, Rhoads JM. Safety and tolerability of Lactobacillus reuteri DSM 17938 and effects on biomarkers in healthy adults: results from a randomized masked trial. PLoS One. 2012;7(9):e43910. doi: 10.1371/journal.pone.0043910. Epub 2012 Sep 6. PMID 22970150